CLINICAL TRIAL: NCT04538625
Title: A Phase 3 Multicenter, Randomized, Double-blind Placebo-controlled Trial Evaluating Crofelemer for the Prophylaxis of Diarrhea in Adult Patients With Solid Tumors Receiving Targeted-cancer Therapies With or Without Standard Chemotherapy
Brief Title: Prophylaxis of Diarrhea in Adult Cancer Patients Receiving Targeted Cancer Therapy
Acronym: OnTARGET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Napo Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NP 303-102
Record Dates: First submitted 2020-08-28; First posted 2020-09-04 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2023-11

CONDITIONS: Cancer Therapy-Related Diarrhea; Chemotherapy-related Diarrhea; Adult Solid Tumor; Prophylaxis of Diarrhea; Symptomatic Relief of Diarrhea; Targeted Therapy-related Diarrhea
MeSH Terms: interventions — crofelemer

STUDY DESIGN:
Intervention Model Description: A randomized, placebo controlled, double blind study to evaluate the safety and efficacy of crofelemer in providing prophylaxis of diarrhea in adult patients with solid tumors receiving targeted cancer therapy containing regimens. Diarrhea grading will be done according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE Ver. 5.0).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects randomized to the placebo arm, will receive oral doses of matching placebo tablets twice daily with or without food.
  Interventions: Drug: Placebo
- Crofelemer (Experimental): Subjects randomized to the crofelemer arm, will receive oral doses of crofelemer 125mg delayed-release tablets twice daily with or without food.
  Interventions: Drug: Crofelemer 125 MG [Mytesi]

INTERVENTIONS:
Drug: Crofelemer 125 MG [Mytesi] — Randomized, Double-blind, Placebo-controlled, two arm trial
  Arms: Crofelemer
Drug: Placebo — Matching placebo tablets
  Arms: Placebo

SUMMARY:
A 24-week, (two 12-week stages), randomized, placebo-controlled, double-blind study to evaluate the safety and efficacy of crofelemer in providing prophylaxis of diarrhea in adult patients with solid tumors treated with targeted cancer therapy-containing treatment regimens. Diarrhea grading will be done according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.

Patients will be randomized 1:1 to placebo or crofelemer and will be stratified by the type of targeted cancer therapy and the tumor type. Placebo and/or crofelemer will be dispensed at Visit 1/Day 1 with the concurrent start of the targeted cancer therapy regimen. The initial Stage I double-blind placebo-controlled primary treatment phase will occur over a 12-week period to accommodate approximately 3 cycle chemotherapy cancer treatment dosing-cycles. The Primary and Secondary Endpoints will be analyzed after the last patient last visit (LPLV) of Stage I.

After completing the Stage I double-blind, placebo-controlled primary treatment phase, the subjects will have the option to remain on their assigned treatment arm and reconsented to enter into the Stage II extension phase. Reconsent will be required to enter into Stage II. For subjects who do not reconsent, visit 5 will be the last study visit.

DETAILED DESCRIPTION:
A randomized, placebo controlled, double blind study to evaluate the safety and efficacy of crofelemer in providing prophylaxis of diarrhea in adult patients with solid tumors receiving targeted cancer therapy containing regimens. Diarrhea grading will be done according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE Ver. 5.0).

Randomization will be at a 1:1 ratio with subjects randomized either to crofelemer 125 mg delayed-release tablets or matching placebo tablets administered orally twice daily with or without food. Randomization will be stratified by the type of targeted cancer therapy and by tumor type. Placebo and crofelemer treatment will be initiated concomitantly with the administration of targeted cancer therapy-containing regimens.

The Stage I double-blind placebo-controlled primary treatment phase will be the first 12-week period to accommodate targeted cancer therapy with approximately three (3) cycle chemotherapy regimens (if needed) over the inclusive 12-week period after initiation of crofelemer or placebo treatment in Stage I.

After completing the Stage I treatment phase (12 weeks), and after the LPLV of the primary Stage I treatment phase, the primary and secondary endpoints will be analyzed. The subjects will have the option to remain on their assigned treatment arm and reconsented to enter into the Stage II extension phase. Reconsent will be required to enter into Stage II. For subjects who do not reconsent, Visit 5 will be the last study visit. Subjects who enter into the Stage II extension phase will continue on their originally assigned study treatment commenced at the beginning of Stage I.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients to receive targeted cancer therapy drugs that have a reported an all grade diarrhea incidence of 50% or higher (e.g., tyrosine kinase inhibitors, cdk inhibitors, anti-EGFR, etc., for treatment of solid tumors.

  2. Patients able to provide written informed consent.

  3. Men and women ≥ 18 years of age.

  4. Pathologically and/or radiologically confirmed diagnosis of solid tumors scheduled to receive targeted cancer therapy.

  5. Patients eligible to receive targeted cancer therapy per NCCN (National Comprehensive Cancer Network) guidelines and/or standard-of-care practice, with or without cycle chemotherapy.

  6. Patient can receive concomitant cycle [standard] chemotherapy agents together with their targeted cancer therapy treatment regimens.

  7. ECOG (Eastern Cooperative Oncology Group) performance status 0-2 and expected to survive a 12-week course of targeted therapy with or without chemotherapy

  8. Negative urine pregnancy test at time of informed consent for women of childbearing potential.

Exclusion Criteria:

* 1. Patients receiving any type of immunotherapy including but not limited to immune checkpoint inhibitors that inhibit negative regulatory components of immune response such as cytotoxic T-lymphocyte associated antigen 4 (CTLA-4) and the programmed cell death protein-1 and its ligand (PD1/ PDL1) and IL-2 cancer immunotherapy.

  2. Any cancer therapy for which antidiarrheal (antimotility) medications in the prophylaxis setting is mandatory, including but not limited to patients receiving neratinib and irinotecan.

  3. Ongoing irritable bowel syndrome (IBS) or colitis (including but not limited to ulcerative colitis, Crohn's disease, microscopic colitis, etc.).

  4. Ongoing diarrhea and/or diarrheal episodes within the previous 7 days prior to randomization into the study.

  5. Laxative use within 7 days prior to randomization or a history of constipation requiring the use of laxatives for more than ≥ 30 consecutive days.

  6. Inadequate organ function, which may include, but is not limited to, the following laboratory results within 28 days prior to signing consent: Total bilirubin > upper limit of normal (ULN), AST (SGOT) and ALT (SPGT) > 2.5 ULN (unless the participant has documented Gilbert's syndrome, hepatocellular carcinoma or hepatic metastases), serum creatinine > 2.0 mg/dL or 177 μmol/L.
  1. NOTE: Investigator discretion will determine continued eligibility after randomization occurs, in the event the liver function test results are greater than (>) the proposed upper limit of normal.

     7. Use of other investigational drugs within 4 weeks of signed informed consent or foreseen use during the study.

     8. Use of antibiotics within the past 7 days (up to 2 prophylactic doses of antibiotic for procedures, including but not limited to port placement, is permitted) prior to randomization.

     9. Total colectomy and/or any type of gastrointestinal ostomy.

     10. Major abdominal or pelvic surgery within the past 3 months.

     11. Previous (within 1 month) or planned abdominal and/or pelvic radiation.

     12. Fecal incontinence from ongoing radiation-induced diarrhea or constipation

     13. Active systemic infection requiring ongoing intervention, including but not limited to oral and intravenous antibiotics, anti-fungals, anti-parasitics, and anti-viral drugs.

     14. Inability to comply with study requirements as judged by the Investigator.

     15. Pregnant and/or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Frequency of Number of Loose/watery Stools | For the entire 12-week double-blind placebo-controlled treatment period (The Stage 1 Primary Treatment Phase).
  The frequency of diarrhea as measured by the average number of loose/watery stools per week will be evaluated as a continuous endpoint.

SECONDARY OUTCOMES:
Proportion of Durable, Clinical Responders | Initial 12-week (Stage 1) period of the study.
  Proportion of "durable responders" defined as the proportion of subjects with ≤7 loose and/or watery bowel movements per week for at least 50% of the time over the Stage 1 double-blind placebo-controlled primary treatment period (Stage 1).
Maximum Number of Weekly Loose/Watery Stools | Initial 12-week (Stage 1) period of the study.
  Maximum number of weekly unformed (loose and/or watery) bowel movements from Week 1 through end of Week 12.
Fecal Incontinence | Initial 12-week (Stage 1) period of the study.
  Mean number of fecal incontinence episodes from Week 1 through end of Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Okhuysen, MD, Principal Investigator — M.D. Anderson Cancer Center; Pravin Chaturvedi, PhD, Study Chair — Napo Pharmaceuticals
Locations (52):
- United States (27):
  - Arizona Oncology Associates PC - HAL, Prescott, Arizona
  - Pacific Cancer Medical Center Inc, Anaheim, California
  - The Oncology Institute of Hope and Innovation, Corona, California
  - The Oncology Institute of Hope and Innovation, Glendale, California
  - PIH Health Whittier Hospital, Whittier, California
  - SCL Health Research Institute, Lafayette, Colorado
  - GenesisCare USA, Aventura, Florida
  - Cancer Care Centers of Brevard, Inc., Palm Bay, Florida
  - BRCR Global, Plantation, Florida
  - Advanced Research Institute, St. Petersburg, Florida
  - American Oncology Partners of Maryland, Bethesda, Maryland
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - North Shore Hematology Oncology Associates dba New York Cancer and Blood Specialists, Port Jefferson Station, New York
  - Jacobi Medical Center, The Bronx, New York
  - Gabrail Cancer Research, Canton, Ohio
  - Oregon Health & Science University (OHSU) Knight Cancer Institute, Portland, Oregon
  - The West Clinic Research, Germantown, Tennessee
  - Texas Oncology - Denison, Denison, Texas
  - Texas Oncology, P.A. - Flower Mound, Flower Mound, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - New Braunfels, New Braunfels, Texas
  - Texas Oncology - Plano East, Plano, Texas
  - Texas Oncology - Gulf Coast, Webster, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Shenandoah Oncology Associates, Winchester, Virginia
  - MultiCare Institute for Research and Innovation, Tacoma, Washington
- Argentina (8):
  - Fleischer Medical Center, Buenos Aires
  - Medical Center Austral, Buenos Aires
  - Buenos Aires British Hospital, Buenos Aires
  - Cordoba Oncology Institute (IONC), Córdoba
  - Center of Nuclear and Molecular Medicine of Entre Rios (CEMENER), Paraná
  - CEDIT Diagnostic and Treatment Center, Salta
  - 9 of July Sanatorium, San Miguel de Tucumán
  - Isis Specialized Clinic, Santa Fe
- Georgia (5):
  - LLC "Todua Clinic", Tbilisi
  - Archangel St. Michael Multiprofile Clinical Hospital LTD, Tbilisi
  - JSC K. Eristavi National Center of Experimental and Clinical Surgery, Tbilisi
  - Malkhaz Katsiashvili Multiprofile Emergency Medicine Center LLC, Tbilisi
  - LTD Caucasus Medical Centre, Tbilisi
- Serbia (6):
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - National Cancer Research Center, Belgrade
  - Institute of Pulmonary Diseases of Vojvodina, Kamenitz
  - Oncology Institute of Vojvodina (IOV), Kamenitz
  - University Clinical Center Kragujevac, Kragujevac
  - University Clinical Center Nis, Niš
- Taiwan (6):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chi Mei Medical Center - LiouYing Branch, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hirsh V, Blais N, Burkes R, Verma S, Croitoru K. Management of diarrhea induced by epidermal growth factor receptor tyrosine kinase inhibitors. Curr Oncol. 2014 Dec;21(6):329-36. doi: 10.3747/co.21.2241. PMID 25489260
- [Background] Davila M, Bresalier RS. Gastrointestinal complications of oncologic therapy. Nat Clin Pract Gastroenterol Hepatol. 2008 Dec;5(12):682-96. doi: 10.1038/ncpgasthep1277. Epub 2008 Oct 21. PMID 18941434
- [Background] Gibson RJ, Keefe DM. Cancer chemotherapy-induced diarrhoea and constipation: mechanisms of damage and prevention strategies. Support Care Cancer. 2006 Sep;14(9):890-900. doi: 10.1007/s00520-006-0040-y. Epub 2006 Apr 8. PMID 16604351
- [Background] Stein A, Voigt W, Jordan K. Chemotherapy-induced diarrhea: pathophysiology, frequency and guideline-based management. Ther Adv Med Oncol. 2010 Jan;2(1):51-63. doi: 10.1177/1758834009355164. PMID 21789126
- [Background] Engelking C, Rutledge DN, Ippoliti C, Neumann J, Hogan CM. Cancer-related diarrhea: a neglected cause of cancer-related symptom distress. Oncol Nurs Forum. 1998 Jun;25(5):859-60. No abstract available. PMID 9644701
- [Background] Benson AB 3rd, Ajani JA, Catalano RB, Engelking C, Kornblau SM, Martenson JA Jr, McCallum R, Mitchell EP, O'Dorisio TM, Vokes EE, Wadler S. Recommended guidelines for the treatment of cancer treatment-induced diarrhea. J Clin Oncol. 2004 Jul 15;22(14):2918-26. doi: 10.1200/JCO.2004.04.132. PMID 15254061
- [Background] Di Fiore F, Van Cutsem E. Acute and long-term gastrointestinal consequences of chemotherapy. Best Pract Res Clin Gastroenterol. 2009;23(1):113-24. doi: 10.1016/j.bpg.2008.11.016. PMID 19258191
- [Background] Carlotto A, Hogsett VL, Maiorini EM, Razulis JG, Sonis ST. The economic burden of toxicities associated with cancer treatment: review of the literature and analysis of nausea and vomiting, diarrhoea, oral mucositis and fatigue. Pharmacoeconomics. 2013 Sep;31(9):753-66. doi: 10.1007/s40273-013-0081-2. PMID 23963867
- [Background] Bowen JM. Mechanisms of TKI-induced diarrhea in cancer patients. Curr Opin Support Palliat Care. 2013 Jun;7(2):162-7. doi: 10.1097/SPC.0b013e32835ec861. PMID 23399616
- [Background] Crutchley RD, Miller J, Garey KW. Crofelemer, a novel agent for treatment of secretory diarrhea. Ann Pharmacother. 2010 May;44(5):878-84. doi: 10.1345/aph.1M658. Epub 2010 Apr 13. PMID 20388859
- [Background] Cottreau J, Tucker A, Crutchley R, Garey KW. Crofelemer for the treatment of secretory diarrhea. Expert Rev Gastroenterol Hepatol. 2012 Feb;6(1):17-23. doi: 10.1586/egh.11.87. PMID 22149578
- [Background] Tradtrantip L, Namkung W, Verkman AS. Crofelemer, an antisecretory antidiarrheal proanthocyanidin oligomer extracted from Croton lechleri, targets two distinct intestinal chloride channels. Mol Pharmacol. 2010 Jan;77(1):69-78. doi: 10.1124/mol.109.061051. Epub 2009 Oct 6. PMID 19808995
- [Background] Holodniy M, Koch J, Mistal M, Schmidt JM, Khandwala A, Pennington JE, Porter SB. A double blind, randomized, placebo-controlled phase II study to assess the safety and efficacy of orally administered SP-303 for the symptomatic treatment of diarrhea in patients with AIDS. Am J Gastroenterol. 1999 Nov;94(11):3267-73. doi: 10.1111/j.1572-0241.1999.01535.x. PMID 10566728
- [Background] DiCesare D, DuPont HL, Mathewson JJ, Ashley D, Martinez-Sandoval F, Pennington JE, Porter SB. A double blind, randomized, placebo-controlled study of SP-303 (Provir) in the symptomatic treatment of acute diarrhea among travelers to Jamaica and Mexico. Am J Gastroenterol. 2002 Oct;97(10):2585-8. doi: 10.1111/j.1572-0241.2002.06027.x. PMID 12385443
- [Background] Mangel AW, Chaturvedi P. Evaluation of crofelemer in the treatment of diarrhea-predominant irritable bowel syndrome patients. Digestion. 2008;78(4):180-6. doi: 10.1159/000185719. Epub 2008 Dec 18. PMID 19092244
- [Background] Pessi MA, Zilembo N, Haspinger ER, Molino L, Di Cosimo S, Garassino M, Ripamonti CI. Targeted therapy-induced diarrhea: A review of the literature. Crit Rev Oncol Hematol. 2014 May;90(2):165-79. doi: 10.1016/j.critrevonc.2013.11.008. Epub 2013 Dec 5. PMID 24373918
- [Background] Macarthur RD, Hawkins TN, Brown SJ, Lamarca A, Clay PG, Barrett AC, Bortey E, Paterson C, Golden PL, Forbes WP. Efficacy and safety of crofelemer for noninfectious diarrhea in HIV-seropositive individuals (ADVENT trial): a randomized, double-blind, placebo-controlled, two-stage study. HIV Clin Trials. 2013 Nov-Dec;14(6):261-73. doi: 10.1310/hct1406-261. PMID 24334179
- [Background] Nee J, Salley K, Ludwig AG, Sommers T, Ballou S, Takazawa E, Duehren S, Singh P, Iturrino J, Katon J, Lee HN, Rangan V, Lembo AJ. Randomized Clinical Trial: Crofelemer Treatment in Women With Diarrhea-Predominant Irritable Bowel Syndrome. Clin Transl Gastroenterol. 2019 Dec;10(12):e00110. doi: 10.14309/ctg.0000000000000110. PMID 31800542